CLINICAL TRIAL: NCT06291272
Title: Randomised Placebo Controlled Trial of Methylcellulose or Psyllium on Fermentation of inUlin Assessed USing MRI (RUFUS)
Brief Title: Effect of Methylcellulose or Psyllium on Fermentation of inUlin Assessed USing MRI
Acronym: RUFUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FMHS 328-0723
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Colon, Irritable
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Psyllium; Methylcellulose; Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: 3 way cross -over
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Opaque plastic bags containing test meals prepared by some one not involved in analysis pf results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psyllium (Experimental): 375 ml containing 15g inulin made up in 375 ml water with 15 g psyllium husk
  Interventions: Dietary Supplement: Psyllium; Dietary Supplement: Inulin
- Methylcelulose (Experimental): 375 ml containing 15g inulin made up in 375 ml water with 15g modified methylcellulose
  Interventions: Dietary Supplement: Methylcellulose; Dietary Supplement: Inulin
- Maltodextrin (Placebo Comparator): 375 ml containing 15g inulin made up in 375 ml water with maltodextrin powder (placebo)
  Interventions: Dietary Supplement: Inulin; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Psyllium — 15 g psyllium + 15 g inulin
  Arms: Psyllium
Dietary Supplement: Methylcellulose — 15 g methylcellulose + 15 g inulin
  Arms: Methylcelulose
Dietary Supplement: Inulin — 15 inulin
Dietary Supplement: Maltodextrin — 15 maltodextrin
  Arms: Maltodextrin

SUMMARY:
The challenge is to understand how fibre interacts with whole-gut function to alter colonic fermentation of fermentable oligo-di- and mono-saccharides and polyhydric alcohols (FODMAPs). Studies will exploit the recent availability of a range of food grade modified celluloses which can form gels at body temperature to perform human studies to explore whether the beneficial effect of psyllium is unique or will be found with all gelling substances (4). The investigators are currently performing the COCOA2 study (Effect of modified cellulose on colonic fermentation of inulin) using a modified methylcellulose (results awaited). The investigators now wish to image what happens in the colon when methylcellulose is ingested to enable planning of the next step in the research programme.

DETAILED DESCRIPTION:
Aim The aim is to test the hypothesis that a gel of either methylcellulose or psyllium incorporating inulin will reduce colonic gas volumes assessed by MRI 0-6 hours and 24 hours post ingestion as compared to inulin combined with placebo, maltodextrin.

Objective The primary objective is to define the effect of methylcellulose and /or psyllium on colonic gas as assessed by MRI. Previous studies have used large doses to ensure a large effect to avoid a type II error however the doses used are well outside the normal consumption. The investigators wish to compare the effect of the methylcellulose mix on the fermentation of 15 g of inulin.

Secondary Objectives A) Assess the effect of methylcellulose on gastric emptying, oro-cecal transit time (OCTT) by MRI assessment of arrival of "head of meal", regional MRI colonic appearances, including signal intensity at 6 and 24 hours to determine the likely length of effect, C) to asses breath hydrogen production over 24 hour post ingestion including overnight assessments, D) to assess Whole Gut Transit Time (WGTT) using blue muffins test, E) to measure AUC (0-24) for breath methane; F) to measure gas production over 48 hours incubation in vitro model of colon (in collaboration with Quadram Institute); G) to measure metabolite production (short chain fatty acids) using in vitro model of colon(in collaboration with Quadram Institute); H) to analyse microbiota using 16sRNA gene (in collaboration with Quadram Institute); I) to assess the effect of habitual dietary FODMAPs intake on breath hydrogen response to inulin.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent.
* Scoring ≤5 (i.e., mild, or less) for symptoms of flatulence, bloating, abdominal pain, loose stool, and hard stool in previous 2 weeks using a modified Gastrointestinal Symptom Rating Scale (5).
* Agrees to consume the meals provided.
* Agrees to not smoke during the breath hydrogen sampling period.

Exclusion Criteria:

* • Pregnancy, lactating, or planning pregnancy during the course of the investigation declared by candidate.

  * History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function.
  * Reported history of previous resection of the oesophagus, stomach, or intestine (excluding appendix).
  * Intestinal stoma.
  * Have contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury.
  * Unable to lie flat and relatively still for less than 5 minutes.
  * Any medical condition making participation potentially compromising participation in the study e.g., diabetes mellitus, respiratory disease limiting ability to use breath hydrogen analyser, known intolerance to one of the test substances.
  * Has a body mass index (BMI) value less than 18.5 or greater than 35.
  * Will not agree to follow dietary and lifestyle restrictions required.
  * Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors, low dose tricyclic antidepressants, antihistamines, and oral contraceptive pill will be recorded in the CRF but will not be an exclusion criteria).
  * Participants who are taking antibiotics or probiotics as it might alters gut microbiota.
  * Poor understanding of English language.
  * Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM.
  * Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g., cognitive dysfunction, chaotic lifestyle related to substance abuse.
  * Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
colonic gas volume | 0-6 hours
  AUC 0-6 hours of colonic gas volume

SECONDARY OUTCOMES:
colonic gas volume at 6 hours | 0-6 hours
  MRI assessed colonic gas volume at 6 hours
Breath hydrogen | 0-6 hours
  Area under curve (AUC) from time 0-6 hours of breath hydrogen (ppm.hours)
Oro-cecal transit time | 0- 6 hours
24 hour breath hydrogen | 0-24 hours
  Area under curve (AUC) from time 0-24 hours of breath hydrogen (ppm.hours)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MD, Principal Investigator — Professor
Locations (1):
- Nottingham Digestive Disease Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No